CLINICAL TRIAL: NCT05880719
Title: Pilot and Descriptive Study of the Effects of the Implementation of Computer Assisted Music Remediation Groups on the Cognitive Functioning of Young Patients Presenting a First Episode Psychosis
Brief Title: Pilot and Descriptive Study of the Effects of Setting up Computer-assisted Music (CAM) Remediation Groups on the Cognitive Functioning of Young Patients With a First Episode Psychosis (PEP)
Acronym: MAOPEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0179
Record Dates: First submitted 2022-05-31; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Psychotic Episode
Keywords: Music; Computer Aided Music; Memory; First Psychotic Episode

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer-assisted music remediation groupe (Experimental): All participants benefit from 10 sessions of computer-assisted music remediation.These 10 sessions are spread over 3 month every Week.
  Interventions: Other: Computer-assisted Music remediation

INTERVENTIONS:
Other: Computer-assisted Music remediation — These sessions of computer-assisted music remediation last 1h and are each divide in 4 parts :
  * 15 minutes of music improvisation
  * 20 minutes of harmony and rythm exercices
  * 20 minutes of Lesson about the software and musical interfaces
  * 5 minutes of debrief.

SUMMARY:
The use of music in the field of cognitive remediation is growing and much research has focused on the relevance and effectiveness of its use in care. Studies have therefore made it possible to show the relevance of the use of musical material in the remediation of patients with various pathologies with cognitive disorders (head trauma, stroke, Alzheimer's disease). Although cognitive remediation has been widely studied in patients with schizophrenia, few studies suggest the effects of remediation in patients with a first psychotic episode. No study currently demonstrates the relevance of this material in the remediation of young people presenting a first psychotic episode.

The Mobile Intensive Care Team of the Adult Psychiatry Service of the CHU de Caen (EMSI) takes care of patients who have presented with a first psychotic episode. Young people entering an emerging psychosis frequently exhibit cognitive impairment. These attacks are variable and can concern memory, attentional and executive functioning. The most frequent disorders concern memory functioning and it is important to deal with them early in order to improve the functional prognosis of the young person.

We therefore propose the establishment of cognitive remediation groups through the MAO with patients treated by EMSI. These groups would aim to heal memory, attention and executive functions through exercises and musical practice through the Ableton © software. We therefore propose a study that would assess the effects of these workshops on the cognitive functioning of patients with memory difficulties. Attentional and executive functioning as well as self-esteem and negative symptoms will also be assessed.

This remedy will be offered in groups of 4. In this feasibility study, 30 patients will be included depending on the inclusion and monitoring capacities of the center. Ten weekly sessions of one hour per group over a period of 3 months will be applied. To assess the beneficial effects of this group remediation, assessments will be carried out at the start of the study and at the end of the 10 sessions.

The aim of this study is to assess the effects of an CAM remediation group on cognitive functioning, mood and self-esteem in patients who presented with a first psychotic episode.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 30 years.
* Consult for a first psychotic episode according to the criteria of the DSM-V
* Francophone patient
* With at least one memory deficit highlighted at the neuropsychological assessment of entry into the EMSI
* Benefiting from a follow-up within the EMSI
* Affiliated to the social security system
* Clinically stabilized patient one month away from psychiatric hospitalization
* Patient who has been informed of the study and has given his informed consent.

Exclusion Criteria:

Inability to give the patient informed information

* Not meeting the criteria of the DSM-V of first episode of psychosis
* Absence of memory cognitive disorders at the neuropsychological assessment of entry into the EMSI department.
* Patient who has already had cognitive remediation in his EMSI management.
* Patients under judicial protection measure (guardianship or curatorship).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
A statistical significant change in episodic memory functionning from Baseline 1 to Baseline 2 (Week 14). | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the episodic verbal memory will be performed at Baseline 1 (Week 0) and at Baseline 2 (Week 14) with the WMS-IV (Weschler Memory Scale 4th edition). This scale provides an episodic memory measure varying from 60 to 140 (mean = 100 ; standard deviation = 15). This measure is called Delayed Memory Index.

SECONDARY OUTCOMES:
A statistical significant change in working memory functionning from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the episodic verbal memory will be performed at Baseline 1 and at Baseline 2 with the WMS-IV (Wechsler Memory Scale 4th edition). This scale provides a working memory measure varying from 60 to 140 (mean = 100; standard deviation = 15). This measure is called Immediate Memory Index.
A statistical significant change in mental flexibility from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the mental flexibility will be performed at Baseline 1 and at Baseline 2 with de Modified Card Sorting Test. This test provides a mental flexibility measure using the errors numbers at the task.
A statistical significant change in mental flexibility from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the mental flexibility will be performed at Baseline 1 and at Baseline 2 with the verbal fluency test. This test provides a mental flexibility measure using the number of words given through 2 minutes.
A statistical significant change in inhibition ability from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessement of the inhibition ability will be performed at Baseline 1 and Baseline 2 with the Stroop test. This test provides an inhibition measure using the errors numbers at this task.
A statistical significant change in sustained attention ability from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the sustained attention will be performed at Baseline 1 and Baseline 2 with the PASAT (Paced Auditory Serial Addition Test ). This test provides an sustained attention measure using an overall score.
A statistical significant change in processing speed from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the processing speed will be performed at Baseline 1 and Baseline 2 with the symbols subtest of the WAIS-IV (Wechsler Adult Intelligence Scale 4th edition). This test provides a processing speed measure using an overall score.
A statistical significant change in humor from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the humor will be performed at Baseline 1 and Baseline 2 with the Calgary scale. This scale provides an humor overall score varying from 0 to 27. Above the treshold score of 6 there is a major depressive episode.
A statistical significant change in self-esteem from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the self-esteem will be performed at Baseline 1 and Baseline 2 with the SERS (Self-Esteem Rating Scale). This scale gives a self-esteem measure using two overall score from -70 to -10 and from 10 to 70 according to the scales.
A symptomatology statistical significant change from Baseline 1 to Baseline 2. | Baseline 1 (Week 0) and Baseline 2 (Week 14)
  An assessment of the symptomatology will be performed at Baseline 1 and Baseline 2 with the PANSS (Positive And Negative Syndrom Scale). This scale provides an overall score varying from 40 to 280. A higher score means importants symptômes.

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France